CLINICAL TRIAL: NCT01483872
Title: Phase II Trial of a Novel Catheter Lock Solution For Adjunctive Treatment of Hemodialysis Catheter-Associated Bacteremia.
Brief Title: Use of a Novel Catheter Lock Solution For Treatment of Hemodialysis Catheter Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to poor enrollment.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Saima Aslam, Asst Adjunct Prof, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101094
Record Dates: First submitted 2011-11-26; First posted 2011-12-02 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Infection; Dialysis Catheter
Keywords: salvage infected hemodialysis catheters; novel catheter lock solution
MeSH Terms: conditions — Infections | interventions — Heparin; Citric Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAC/Tigecycline/Heparin combination lock solution (Experimental): A combination of the above three drugs will form the catheter lock solution that will be instilled into the catheter
  Interventions: Drug: NAC/Tigecycline/Heparin combination lock solution
- Standard anticoagulant (heparin or citrate) (Placebo Comparator): Standard anticoagulant (heparin or citrate)
  Interventions: Drug: Standard anticoagulant (Heparin or Citrate)

INTERVENTIONS:
Drug: NAC/Tigecycline/Heparin combination lock solution
  Arms: NAC/Tigecycline/Heparin combination lock solution
Drug: Standard anticoagulant (Heparin or Citrate)
  Arms: Standard anticoagulant (heparin or citrate)

SUMMARY:
Aim: To conduct a randomized, double-blinded, controlled phase II trial to investigate the use of a catheter lock solution consisting of N-acetylcysteine, tigecycline and heparin, in addition to systemic antibiotics, for the treatment of hemodialysis catheter-associated bacteremia via a catheter-salvage strategy.

The investigators plan to randomize 102 patients with hemodialysis catheter-associated bacteremia to one of two treatment arms. All patients will receive systemic antibiotics for treatment of their infection. Additionally, patients randomized to the interventional arm will also receive a catheter lock solution consisting of N-acetylcysteine, tigecycline and heparin for 2 weeks with the aim of salvaging the catheter. The control arm will receive only an anticoagulant solution as a catheter lock which is standard of care - this can be either heparin or citrate (depending on what agent is standard of care for a particular patient). The main outcome of interest is successful treatment which is defined as a resolution of the current episode of bacteremia as well as lack of recurrent bacteremia within 90 days of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (≥ 18 years of age) who has ESRD and a prevalent or incident tunneled hemodialysis catheter and expected to continue hemodialysis for 3 months will be eligible for enrollment.

Exclusion Criteria:

* The following patients will be excluded from study entry:

  1. patient is unable (and no guardian or legal representative is available) or unwilling to provide informed consent and
  2. patient is allergic to NAC, tigecycline, minocycline, or heparin.

The following patients will be excluded from randomization:

1. patient has evidence of a complicated bacteremia such as endocarditis, septic thrombophlebitis, septic emboli, osteomyelitis, deep seated abscess, or hypotension requiring use of vasopressors,
2. patient has evidence of an exit site infection around the catheter such as a pus pocket, purulent drainage, or erythema,
3. patient is pregnant or will become pregnant,
4. the infection is due to an organism that is resistant to tigecycline such as Candida or Pseudomonas species.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Medical Center, San Diego, California, United States

REFERENCES:
- [Derived] Almeida BM, Moreno DH, Vasconcelos V, Cacione DG. Interventions for treating catheter-related bloodstream infections in people receiving maintenance haemodialysis. Cochrane Database Syst Rev. 2022 Apr 1;4(4):CD013554. doi: 10.1002/14651858.CD013554.pub2. PMID 35363884

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 patients signed consent forms. Only one developed an active infection and thus underwent randomization.
Groups:
- NAC/Tigecycline/Heparin Combination Lock Solution: A combination of the above three drugs will form the catheter lock solution that will be instilled into the catheter
  NAC/Tigecycline/Heparin combination lock solution
Period: Overall Study
Arm/Group | NAC/Tigecycline/Heparin Combination Lock Solution | Standard Anticoagulant (Heparin or Citrate)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Nine participants signed consent forms, only one randomized. Data was not analyzed.
Time Frame: 90 days
Population: Nine participants signed consent forms, only one randomized. Data was not analyzed.
Groups:
- All Participants: Nine participants signed consent forms, only one randomized. Data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Nine participants signed consent forms, only one randomized. Study terminated due to low enrollment. Data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes